CLINICAL TRIAL: NCT00144482
Title: A Randomized, Double-Blind Study of Recombinant Human Erythropoietin in Anemic Cancer Patients Undergoing Chemotherapy
Brief Title: A Study of Recombinant Human Erythropoietin in Anemic Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPO307JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Chemotherapy Induced Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: recombinant human erythropoietin
- 2 (Placebo Comparator)
  Interventions: Drug: recombinant human erythropoietin placebo

INTERVENTIONS:
Drug: recombinant human erythropoietin — 36000IU（0.5mL）s.c./week for 8 weeks
  Arms: 1
Drug: recombinant human erythropoietin placebo — 0 IU(0.5mL)s.c./week for 8 weeks
  Arms: 2

SUMMARY:
To evaluate the effectiveness and safety in randomized, double-blind, parallel-group study in anemic cancer patients undergoing chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients

Exclusion Criteria:

* a history of myocardial, cerebral or pulmonary infarction
* severe hypertension beyond control by drugs

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2003-12; Primary Completion 2005-03 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
The increase in Hb concentration | week 8

SECONDARY OUTCOMES:
Changes in QOL scores | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiharu Ishikura, Study Director — Chugai Pharmaceutical